CLINICAL TRIAL: NCT04683692
Title: A Pilot Randomized Study of the Use of The Sentinel Device for Cerebral Protection During Atrial Fibrillation Ablation: MRI Imaging and Laboratory Sub-study
Brief Title: A Study to Assess the Use of The Sentinel Device During Atrial Fibrillation Ablation
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: This sub-study was combined to the parent study protocol (NCT04685317)
Sponsor: Mayo Clinic (Other)
Collaborators: Boston Scientific Corporation (Industry)
Responsible Party: Principal Investigator, Ammar M. Killu, Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 20-001308
Record Dates: First submitted 2020-09-25; First posted 2020-12-24 (Actual); Last update posted 2023-04-14 (Actual); Status verified 2023-04

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation | interventions — Magnetic Resonance Imaging

STUDY DESIGN:
Intervention Model Description: Parent Study Design: Patients undergoing clinically indicated catheter ablation for AF in the parent study will be randomized 2:1 to two arms: (1) cerebral protection with the Sentinel device and (2) control group without cerebral protection
Masking Description: For both the parent study and the sub-study, participants and investigators will be unblinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Cerebral protection with the Sentinel device (Experimental): Subjects who received the Sentinel device in the parent study
  Interventions: Device: Magnetic Resonance Imaging (MRI); Other: Laboratory Testing
- Control group without cerebral protection (Active Comparator): Subjects who did not received the Sentinel device in the parent study
  Interventions: Device: Magnetic Resonance Imaging (MRI); Other: Laboratory Testing

INTERVENTIONS:
Device: Magnetic Resonance Imaging (MRI) — Cerebral MRI will be performed without gadolinium contrast using a 3 Tesla scanner prior to and 1 to 7 days after catheter ablation
Other: Laboratory Testing — Laboratory blood testing to include high sensitivity CRP (hs-CRP), interleukin-6 (IL-6), NT-proBNP and high sensitivity troponin prior to and post-ablation

SUMMARY:
Researchers are determining whether the use of the Sentinel cerebral protection device during atrial fibrillation ablation will affect the occurrence of new cerebral infarcts in brain MRI. We are also studying if laboratory tests can be used to predict the rate of cerebral infarction and microbleeds in patients undergoing atrial fibrillation (AF) ablation procedures with and without use of the Sentinel Device.

DETAILED DESCRIPTION:
Patients currently participating in the research study titled: "A Pilot Randomized Study of the Use of the Sentinel Device for Cerebral Protection during Atrial Fibrillation Ablation" will be asked to participate in this sub-study to collect additional MRI and laboratory data to support the main study. This study will assess the number, size and volume of new cerebral emboli in protected territories detected using MRI of the brain within 7 days after AF ablation in patients treated with the Sentinel device compared to controls not receiving the Sentinel device, and to assess if change in blood inflammatory markers is associated with silent cerebral lesions.

ELIGIBILITY:
Inclusion Criteria:

* Patients over the age of 18 years undergoing radiofrequency or cryoballoon ablation for AF who provide informed consent will be included

Exclusion Criteria:

* Severe peripheral arterial disease that precludes deployment of Sentinel device
* Unable to undergo MRI brain due to the presence of an MRI noncompatible implanted device
* Unable or unwilling to provide informed consent.
* Known history of dementia.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-03 (Estimated); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
New cerebral infarcts | day 1 to 7 after atrial fibrillation ablation
  Total number of new cerebral infarcts in the protected territories detected on brain MRI after ablation in the Sentinel device group vs control group
Change in high sensitivity CRP (hs-CRP) | baseline 1 - 30 days prior to ablation, days 1 - 7 after atrial fibrillation ablation
  High sensitivity CRP (hs-CRP) measured in mg/L to detect changes in peripheral markers of inflammation
Change in interleukin-6 (IL-6) | baseline 1 - 30 days prior to ablation, days 1 - 7 after atrial fibrillation ablation
  Interleukin-6 measured in pg/ml to detect changes in peripheral markers of inflammation
Change in NT-proBNP | baseline 1 - 30 days prior to ablation, days 1 - 7 after atrial fibrillation ablation
  NT-proBNP measured in pg/ml to detect changes in tissue damage
Change in high sensitivity troponin | baseline 1 - 30 days prior to ablation, days 1 - 7 after atrial fibrillation ablation
  High sensitivity troponin measure in ng/mL to detect changes in tissue damage

CONTACTS AND LOCATIONS:
Overall Officials: Ammar Killu, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials